CLINICAL TRIAL: NCT06398457
Title: A Pilot Study of Darzalex Faspro (Daratumumab and Hyaluronidase-fihj) Before Standard Desensitization and Allogeneic Peripheral Blood Stem Cell Transplantation in Adult Patients at High-risk for Primary Graft Failure Secondary to Donor Specific Antibodies
Brief Title: Darzalex Faspro (Daratumumab and Hyaluronidase-fihj) Before Standard Desensitization and Allogeneic Peripheral Blood Stem Cell Transplantation in Adult Patients at High-risk for Primary Graft Failure Secondary to Donor Specific Antibodies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2450; IRB00440881 (Other: JHM IRB)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy; Bone Marrow Transplant Rejection; Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS); Acute Lymphoblastic Leukemia (ALL), Adult; Multiple Myeloma; Aplastic Anemia; Lymphoma; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Chronic Myeloid Leukemia; Myelofibrosis
Keywords: DSA; donor specific antibodies; desensitization; BMT; allogeneic stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Anemia, Aplastic; Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Daratumumab-SC (days -42, -35, -28, -21) followed by standard of care DSA desensitization and alloBMT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Daratumumab-SC followed by standard of care DSA desensitization and alloBMT (Experimental): Darzalex Faspro (Daratumumab and hyaluronidase-fihj) will be administered subcutaneously (SC) weekly (every 7 day +/- 1 day) for a total of four doses followed by standard desensitization regimen and allogeneic stem cell transplant.
  Interventions: Drug: Darzalex Faspro (Daratumumab and hyaluronidase-fihj); Device: JH-DSA Semi-Quant Screen and Response Score

INTERVENTIONS:
Drug: Darzalex Faspro (Daratumumab and hyaluronidase-fihj) — Darzalex Faspro will be administered weekly as a subcutaneous injection on Days -42, -35, -28 and -21 (+/- 1 day) for a total of four doses at 1800 mg each.
Device: JH-DSA Semi-Quant Screen and Response Score — Serum based semi-quantifiable investigational testing regimen used to screen for high DSA level or assess response to desensitization. It is based on results from cross-matched flow cytometric assessment cellular-based and solid phase immunoassays (SPI) that estimates antibody level.
  Other Names: JH-DSA Semi-Quant Screen Score; JH-DSA Semi-Quant Response Score

SUMMARY:
This research is being done to investigate the safety and effectiveness of Darzalex Faspro (daratumumab and hyaluronidase-fihj) (a monoclonal antibody that targets plasma cells that make antibodies) and whether it can lower donor specific antibodies (DSA) levels to low enough levels to permit patients to proceed with allogeneic peripheral blood transplant (alloBMT). Those being asked to participate have high DSA levels that puts those being asked to participate at high risk of rejecting the available donor's blood stem cells and making those being asked to participate ineligible to receive a stem cell transplant.

DETAILED DESCRIPTION:
Allogeneic blood or bone marrow transplant (alloBMT) remains the definitive curative treatment for many with relapsed or refractory hematologic malignancies. In recent years, increased use of alternative (non-fully human leukocyte antigen (HLA)-matched) donors has led to increased rates of donor specific antibodies (DSA). DSA are pre-formed HLA-antibodies in the recipient directed against the donor's class I and/or class II HLA antigens. DSA can be formed by exposure to foreign HLA antigens most commonly by pregnancy, blood transfusions, and previous organ or blood transplantation.

High levels of circulating anti-HLA antibodies directed towards mismatched donor HLA antigens at the time of alloBMT can dramatically increase the risk of primary graft failure (PGF). The strength of these donor specific antibodies (DSA) can be assessed with several methodologies including cross-matched cellular based assays (cytotoxic or flow cytometric assessment) or the more sensitive solid phase immunoassay (SPI) that estimates antibody level. Methods to "desensitize" patients with elevated DSAs using therapeutic plasma exchange (TPE), intravenous immunoglobulin (IVIG), and immunosuppression (i.e., mycophenolate mofetil and tacrolimus) are successful in patients with moderate levels of DSAs. However, in many patients, the DSA levels are considered too high for desensitization, or, desensitization has failed to lower levels of the DSA, and suitable alternative donors cannot be readily identified.

In this single-institution study at the Johns Hopkins Sidney Kimmel Comprehensive Cancer Center (SKCCC), we will identify patients in whom alloBMT is indicated, but where DSA levels are above a pre-defined threshold using a proprietary algorithm that combines information from flow cytometric crossmatch (FCXM) and SPI (the Johns Hopkins (JH)-DSA Semi-Quant Screen Score). Patients who meet eligibility criteria will undergo 4 weekly doses of treatment with Darzalex Faspro, an anti- 38 (cluster of differentiation 38) antibody that kills plasma cells and lowers immunoglobulin levels, followed by standard desensitization with TPE, IVIG, and immunosuppression. Eight subjects will be treated in this pilot study. The primary endpoint will be based on safety of Darzalex Faspro and the number of patients who have DSA levels lowered enough to proceed to conditioning based on a pre-defined algorithm called JH-DSA Semi-Quant Response Score.

ELIGIBILITY:
Inclusion Criteria:

1. Participates must meet all other institutional criteria for the planned reduced intensity conditioning allogeneic peripheral blood stem cell transplant (RIC alloHSCT) as defined in Johns Hopkins BMT Policy; all potential non-cord blood donor sources are included: matched related, haploidentical, matched unrelated, mismatched unrelated.
2. Participants must be ≥18 years of age.
3. Participants must have adequate organ function for undergoing RIC allogeneic peripheral blood stem cell transplant, and for undergoing a clinical trial.

   a. Hematologic. i. White blood cell (WBC). ANC ≥ 500/mm3 (growth factor support allowed). ii. Hemoglobin. No specific cut-off. (PRBC transfusion allowed). iii. Platelets. Platelets ≥ 10,000/mm3 (platelet transfusion allowed). b. Liver. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 5x Upper limit of normal (ULN) c. Renal. Serum creatinine ≤ 2.0 mg/dL. d. Cardiac. Left ventricular ejection fraction ≥ 35%. e. Pulmonary. FEV1 ≥ 50%.
4. Subjects are eligible if there are high levels of Donor Specific Antibody levels based on protocol specific scoring system regardless of prior attempts at standard desensitization.
5. Participants must have a no other readily available suitable alternative donor.
6. All potential Participants must be pre-approved by BMT faculty consensus.
7. Participants must have adequate willingness to participate in a clinical trial.

Exclusion Criteria:

1. Previous exposure to Daratumumab-SC or other anti-CD38 therapy

   1. Exposure to Daratumumab-SC or other anti-CD38 therapies (unless a re-treatment study)
   2. Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
   3. Focal radiation therapy within 14 days prior to beginning of planned RIC allogeneic peripheral blood stem cell transplant regimen with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma
2. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
3. Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
4. Known hypersensitivity or intolerance to boron or mannitol, sorbitol, corticosteroids, monoclonal antibodies or human proteins, or the excipients
5. Diagnosis of multiple myeloma or Amyloid light-chain (AL) amyloidosis
6. A planned myeloablative alloBMT or the planned use of bone marrow or cord blood as a stem cell source
7. History of HIV infection at any time in past.
8. Seropositive for hepatitis B (HBV) (defined by a positive test for hepatitis B surface antigen [HBsAg] positive, or antibodies to hepatitis B surface and/or core antigens [antiHBs or antiHBc, respectively] with hepatitis B virus [HBV]- DNA quantitation positive). Patients who are positive for antiHBs and/or antiHBc must have a negative polymerase chain reaction (PCR) for HBV-DNA quantitation result during screening. Patients with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR. Those who are PCR positive will be excluded.
9. Seropositive for hepatitis C (except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy)
10. Clinically significant cardiac disease, including:

    1. Myocardial infarction within 6 months before RIC alloHSCT or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    2. Uncontrolled cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy as assessed by percentage of patients with reduced DSA levels | 2 years
  Efficacy as assessed by the percentage of patients with DSA levels that are reduced to a level permissible for RIC alloHSCT with DSA strength of II or less and at least a 10% decrease in MFI from the baseline as determined by the JH-DSA Response Score.
Safety as assessed by proportion of patients with grade 3 or higher toxicities | 2 years
  Proportion of patients with Grade 3 or higher toxicities attributable to daratumumab for one cycle of Darzalex Faspro

SECONDARY OUTCOMES:
Time (days) to neutrophilic recovery | 2 years
  Average amount of time taken to obtain an absolute neutrophil count (ANC) greater than or equal to 500 (10^6/L) for 3 consecutive days
Time (days) to platelet recovery | 2 years
  Average amount of time taken to reach platelet count greater than 20 (10^9/L) for 3 consecutive days
Number of participants who achieve T-cell chimerism | 2 years
  Number of participants who acheive T cell chimerism by day +60
Number of participants who have primary graft failure | 2 years
  Number of participants who have primary graft failure defined by failure to achieve a T-cell chimerism of 5% or more or neutrophilic engraftment by day +60.

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Gocke, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No